CLINICAL TRIAL: NCT00594542
Title: A Randomized, Double Blind Comparison of the Total Dose of 1.0% Lidocaine With 1:100,000 Epinephrine Versus 0.5% Lidocaine With 1:200,000 Epinephrine Needed to Achieve Effective Anesthesia During Mohs Micrographic Surgery
Brief Title: Comparison of the Total Dose and Efficacy of Two Lidocaine Concentrations Needed for Cutaneous Surgery Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Christopher J. Miller, M.D., University of Pennsylvania Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UPenn IRB-806101
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia
Keywords: lidocaine; local anesthesia; Mohs micrographic surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5% lidocaine group (Experimental): Group that receives 0.5% lidocaine with 1:200,000 epinephrine
  Interventions: Drug: lidocaine
- 1.0% lidocaine group (Experimental): Group that receives 1.0% lidocaine with 1:100,000 epinephrine
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — Each group is the appropriate concentration of lidocaine with epinephrine for local anesthesia at the beginning of each Mohs stage and the reconstruction.

SUMMARY:
The purpose of the study will be to demonstrate whether Mohs micrographic surgery can be performed with a lower total dose of local anesthesia (and greater patient safety) when using 0.5% lidocaine with 1:200,000 epinephrine versus 1% lidocaine with 1:100,000 epinephrine.

DETAILED DESCRIPTION:
The purpose of the study will be to demonstrate whether Mohs micrographic surgery can be performed with a lower total dose of local anesthesia (and greater patient safety) when using 0.5% lidocaine with 1:200,000 epinephrine versus 1% lidocaine with 1:100,000 epinephrine. Mohs micrographic surgery is a multi-staged, same-day procedure used to remove skin cancers under local anesthesia. Reconstruction of the surgical wound is also performed under local anesthesia, usually immediately after achieving tumor clearance.

This randomized, double-blind study will systematically compare the total dose of 1.0% lidocaine with 1:100,000 epinephrine versus 0.5% of lidocaine with 1:200,000 epinephrine needed to achieve local anesthesia during Mohs micrographic surgery (MMS). All healthy adult volunteers (18 years or older) undergoing Mohs micrographic surgery at the Hospital of the University of Pennsylvania's Department of Dermatology and Dermatologic Surgery between June 1, 2007 and August 31, 2007 will be eligible to participate in the study. Our primary intervention will be to record the total dose of lidocaine administered throughout all of the MMS stages and reconstructions using either of the two lidocaine concentrations. A secondary intervention will be to record each patient's level of pain control in order to demonstrate that patient comfort is effectively achieved with a lower total dose of local anesthesia. Pregnant or breast-feeding subjects, those with a history of allergic or other adverse reaction to lidocaine or epinephrine, and those who are cognitively impaired will be excluded. In addition, if the surgeon believes that a patient has a tumor which, due to size or anatomic site, may put him at risk for requiring a dose of lidocaine that approaches the threshold of toxicity, this patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Mohs micrographic surgery patient

Exclusion Criteria:

* Pregnant or breast-feeding subjectsH
* History of allergic or other adverse reaction to lidocaine or epinephrine
* Cognitively impairment
* Surgeon judges patient a risk for lidocaine toxicity due to tumor size

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2007-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a measurement of the total dose of lidocaine (measured in mg) administered to the patient over the course of Mohs micrographic surgery. | One day

SECONDARY OUTCOMES:
The secondary outcome is subject pain, as assessed by a visual analog pain scale and by the volume of extra rescue lidocaine needed during surgery. | One day

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Miller, MD, Principal Investigator — University of Pennsylvania Department of Dermatology